CLINICAL TRIAL: NCT04813796
Title: A Phase 1, Randomized, Observer-Blind, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1283 and mRNA-1273 SARS-CoV-2 Vaccine in Adults Aged 18-55 Years
Brief Title: A Study to Evaluate Safety, Reactogenicity, and Immunogenicity of mRNA-1283 and mRNA-1273 Vaccines in Healthy Adults Between 18 Years and 55 Years of Age to Prevent COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1283-P101
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1283 vaccine; mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants who are offered an opportunity to receive an additional injection of mRNA-1273, will participate in an open-label part of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- mRNA-1283 Dose Level 1 (Experimental): Participants will receive 2 intramuscular (IM) injections of mRNA-1283 at Dose Level 1 on Day 1 and Day 29.
  Interventions: Biological: mRNA-1283
- mRNA-1283 Dose Level 2 (Experimental): Participants will receive 2 IM injections of mRNA-1283 at Dose Level 2 on Day 1 and Day 29.
  Interventions: Biological: mRNA-1283
- mRNA-1283 Dose Level 3 (Experimental): Participants will receive 2 IM injections of mRNA-1283 at Dose Level 3 on Day 1 and Day 29.
  Interventions: Biological: mRNA-1283
- mRNA-1273 (Experimental): Participants will receive 2 IM injections of mRNA-1273 at a pre-specified dose for this study on Day 1 and Day 29.
  Interventions: Biological: mRNA-1273
- Placebo / mRNA-1283 (Experimental): Participants will receive 1 IM injection of study drug-matching placebo on Day 1 and 1 IM injection of mRNA-1283 at a pre-specified dose on Day 29. Participants may be offered an opportunity to receive an additional injection of mRNA-1273 at the pre-specified dose on Open-Label Day 1.
  Interventions: Biological: mRNA-1283; Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1283 — Sterile liquid for injection
  Arms: Placebo / mRNA-1283; mRNA-1283 Dose Level 1; mRNA-1283 Dose Level 2; mRNA-1283 Dose Level 3
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: mRNA-1273
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo / mRNA-1283

SUMMARY:
The primary goal for this study is to evaluate the safety and reactogenicity of 3 dose levels of mRNA-1283 and 1 dose level of mRNA-1273 vaccine given to healthy adults in 2 doses, 28 days apart, and 1 dose level of mRNA-1283 administered as a single dose to healthy adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Understands and agrees to comply with the study procedures and provides written informed consent.
* According to the assessment of the investigator, is in good general health and can comply with study procedures.
* Body mass index (BMI) of 18 kilograms/square meter (kg/m^2) to 35 kg/m^2 (inclusive) at the Screening Visit (Day 0).
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection, agreement to continue adequate contraception or abstinence through 3 months following the second injection, and not currently breastfeeding.

Key Exclusion Criteria:

* Known history of SARS-CoV-2 infection or known exposure to someone with SARS-CoV-2 infection or COVID-19 in the past 30 days.
* Positive serology results for SARS-CoV-2 at the Screening Visit. A negative serological test for SARS-CoV-2, performed on a blood sample obtained at the Screening Visit, is required before a participant can be dosed.
* Travel outside of the United States in the 28 days prior to the Screening Visit (Day 0).
* Prior administration of an investigational, authorized, or licensed CoV (for example, SARS-CoV-2, SARS-CoV, or Middle East Respiratory Syndrome [MERS]-CoV) vaccine, based on medical history interview.
* Current treatment with investigational agents for prophylaxis against COVID-19.
* Recent (within the last 12 months) use of a dermal filler.
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids, 10 milligrams (mg)/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Has received or plans to receive any licensed vaccine 28 days prior to the first injection (Day 1) or plans to receive a licensed vaccine within 28 days before or after any study injection, with the exception of licensed influenza vaccines, which may be received more than 14 days before the first study injection or more than 14 days after the second study injection.
* Receipt of systemic immunoglobulins or blood products within 3 months prior to the Screening Visit (Day 0) or plans for receipt during the study.
* Current use of any inhaled substance (for example, tobacco or cannabis smoke, nicotine vapors).
* History of chronic smoking (1 cigarette a day) within 1 year of the Screening Visit.
* Resides in a nursing home.
* Has donated 450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.
* Participated in an interventional clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 36 (7 days after second dose)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 57 (28 days after second dose)
Number of Participants with Medically-Attended AEs (MAAEs), AE of Special Interest (AESIs), and Serious Adverse Events (SAEs) | Up to Day 394 (1 year after second dose)

SECONDARY OUTCOMES:
Geometric Mean (GM) of SARS-CoV-2 Specific Neutralizing Antibody (nAb) | Day 1, Day 29, Day 36, Day 57, Day 209, and Day 394
GM of SARS-CoV-2-Specific Binding Antibody (bAb) | Day 1, Day 29, Day 36, Day 57, Day 209, and Day 394
Seroconversion as Measured by an Increase of SARS-CoV-2-Specific nAb Titer or bAb Titer | Day 1, Day 29, Day 36, Day 57, Day 209, and Day 394
  Seroconversion measured as defined for the study.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Synexus Clinical Research US Phoenix Southeast, Inc., Chandler, Arizona
  - Optimal Research San Diego, LLC, San Diego, California
  - Optimal Research Melbourne, LLC, Melbourne, Florida
  - Optimal Research Illinois, LLC, Peoria, Illinois
  - Optimal Research Texas, LLC, Austin, Texas

REFERENCES:
- [Derived] Yassini P, Hutchens M, Paila YD, Schoch L, Aunins A, Siangphoe U, Paris R. Interim analysis of a phase 1 randomized clinical trial on the safety and immunogenicity of the mRNA-1283 SARS-CoV-2 vaccine in adults. Hum Vaccin Immunother. 2023 Dec 31;19(1):2190690. doi: 10.1080/21645515.2023.2190690. Epub 2023 Apr 19. PMID 37074202